CLINICAL TRIAL: NCT00062348
Title: B-Uptake In Different Tumours Using The Boron Compounds BSH And BPA
Brief Title: Boronophenylalanine-Fructose Complex (BPA-F) and/or Sodium Borocaptate (BSH) Followed By Surgery in Treating Patients With Thyroid Cancer, Head and Neck Cancer, or Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Masking: None | Purpose: Treatment
Other Study IDs: EORTC-11001; EORTC-11001
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer; Head and Neck Cancer; Metastatic Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; untreated metastatic squamous neck cancer with occult primary; recurrent thyroid cancer; stage IV follicular thyroid cancer; stage IV papillary thyroid cancer; stage IVA colon cancer; stage IVB colon cancer; recurrent colon cancer; adenocarcinoma of the colon; recurrent rectal cancer; stage IVA rectal cancer; stage IVB rectal cancer; adenocarcinoma of the rectum; anaplastic thyroid cancer; insular thyroid cancer; thyroid gland medullary carcinoma; liver metastases; stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I papillary thyroid cancer; stage II papillary thyroid cancer; stage III papillary thyroid cancer; stage I follicular thyroid cancer; stage II follicular thyroid cancer; stage III follicular thyroid cancer; recurrent metastatic squamous neck cancer with occult primary; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; tongue cancer
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Colonic Neoplasms; Rectal Neoplasms; Thyroid Carcinoma, Anaplastic; Carcinoma, Medullary; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — 4-boronophenylalanine-fructose; mercaptoundecahydrododecaborate

INTERVENTIONS:
Drug: boronophenylalanine-fructose complex
Drug: sodium borocaptate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Diagnostic procedures using boronophenylalanine-fructose complex (BPA-F) and/or sodium borocaptate (BSH) to detect the presence of boron in tumor cells may help determine whether patients who have thyroid cancer, head and neck cancer, or liver metastases may benefit from boron neutron capture therapy.

PURPOSE: This phase I trial is studying the side effects of giving BPA-F and/or BSH before surgery to detect boron uptake in tissues of patients with primary, metastatic, or recurrent thyroid cancer, head and neck cancer, or liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify additional solid tumors that may benefit from boron neutron capture therapy.
* Determine the boron concentration in the tumor, surrounding tissues, and blood of patients with operable thyroid cancer, squamous cell cancer of the head and neck, or liver metastases secondary to colorectal adenocarcinoma who receive boronophenylalanine-fructose complex (BPA-F) and/or sodium borocaptate (BSH) before surgical resection.
* Determine the feasibility of using these drugs to obtain a favorable absolute boron-10 concentration in the tumor and optimal tumor-to-blood and tumor-to-healthy tissue boron-10 rates in these patients.
* Determine the qualitative and quantitative toxicity of combined BPA-F and BSH administration in these patients.

OUTLINE: This is a multicenter study. Patients are sequentially assigned to 1 of 3 treatment groups.

* Group I: Patients receive boronophenylalanine-fructose complex (BPA-F) IV over 1 hour. Two hours later, patients undergo surgical resection.
* Group II: Patients receive sodium borocaptate (BSH) IV over 1 hour. Twelve hours later, patients undergo surgical resection.
* Group III: Patients receive BSH IV over 1 hour (administered 12 hours prior to surgery) and BPA-F IV over 1 hour (administered 2 hours prior to surgery). Patients then undergo surgical resection.

During the planned surgery, tissue samples from the tumor and surrounding tissues are collected.

Patients are followed on days 1 and 5 and then at 4 weeks.

PROJECTED ACCRUAL: A maximum of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor of 1 of the following malignant tumor types:

  * Squamous cell cancer of the head and neck
  * Thyroid cancer
  * Liver metastases* secondary to colorectal adenocarcinoma NOTE: *Liver metastases are eligible provided colorectal adenocarcinoma has been histopathologically proven and CT scan/MRI shows metastatic lesions in the liver
* Operable disease for which a surgical excision is planned
* Primary, metastatic, or locally recurrent disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* AST and ALT no greater than 2.5 times ULN
* No other severe liver function impairment

Renal

* Creatinine normal
* BUN normal

Cardiovascular

* No congestive heart failure
* No angina pectoris
* No recent coronary artery disease
* No uncontrolled arrhythmias
* No conduction defects
* No other severe heart disease

Pulmonary

* No severe obstructive or restrictive lung disease

Gastrointestinal

* No severe gastrointestinal disease
* No active peptic ulcer disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing serious mental or organic brain disease (e.g., epilepsy)
* No history of phenylketonuria (only in the case of BPA administration)
* No severe allergic disease requiring continuous medication
* No other concurrent severe disease
* No uncontrolled endocrine disease
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 3 months since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the malignant site

Surgery

* See Disease Characteristics

Other

* Recovered from prior antitumor therapy (excluding alopecia)
* No concurrent anticancer treatment or agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2003-04; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Boron uptake ratio in tumor vs normal tissue

SECONDARY OUTCOMES:
Toxicity measured by NCI-CTC v2.0 up to 28 days after injections

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Sauerwein, MD, PhD, Study Chair — Universitaetsklinikum Essen
Locations (1):
- Universitaetsklinikum Essen, Essen, Germany

REFERENCES:
- [Result] Wittig A, Sheu-Grabellus SY, Collette L, Moss R, Brualla L, Sauerwein W. BPA uptake does not correlate with LAT1 and Ki67 expressions in tumor samples (results of EORTC trial 11001). Appl Radiat Isot. 2011 Dec;69(12):1807-12. doi: 10.1016/j.apradiso.2011.02.018. Epub 2011 Feb 16. PMID 21367608
- [Result] Bendel P, Wittig A, Basilico F, Mauri PL, Sauerwein W. Metabolism of borono-phenylalanine-fructose complex (BPA-fr) and borocaptate sodium (BSH) in cancer patients--results from EORTC trial 11001. J Pharm Biomed Anal. 2010 Jan 5;51(1):284-7. doi: 10.1016/j.jpba.2009.08.018. Epub 2009 Aug 22. PMID 19735988
- [Result] Wittig A, Collette L, Appelman K, Buhrmann S, Jackel MC, Jockel KH, Schmid KW, Ortmann U, Moss R, Sauerwein WAG. EORTC trial 11001: distribution of two 10B-compounds in patients with squamous cell carcinoma of head and neck, a translational research/phase 1 trial. J Cell Mol Med. 2009 Aug;13(8B):1653-1665. doi: 10.1111/j.1582-4934.2009.00856.x. Epub 2009 Jul 10. PMID 19602035
- [Result] Wittig A, Collette L, Moss R, Sauerwein WA. Early clinical trial concept for boron neutron capture therapy: a critical assessment of the EORTC trial 11001. Appl Radiat Isot. 2009 Jul;67(7-8 Suppl):S59-62. doi: 10.1016/j.apradiso.2009.03.012. Epub 2009 Mar 25. PMID 19372041
- [Result] Wittig A, Malago M, Collette L, Huiskamp R, Buhrmann S, Nievaart V, Kaiser GM, Jockel KH, Schmid KW, Ortmann U, Sauerwein WA. Uptake of two 10B-compounds in liver metastases of colorectal adenocarcinoma for extracorporeal irradiation with boron neutron capture therapy (EORTC Trial 11001). Int J Cancer. 2008 Mar 1;122(5):1164-71. doi: 10.1002/ijc.23224. PMID 17985341